CLINICAL TRIAL: NCT05892965
Title: Instant Message-delivered Brief Internet-based Cognitive Behavioural Therapy (iCBT) for Post-stroke Depression: a Mixed Method Study
Brief Title: Instant Message-delivered Brief Internet-based Cognitive Behavioural Therapy (iCBT) for Post-stroke Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 27615721
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Depressive Symptoms; Mobile Phone Use
MeSH Terms: conditions — Stroke; Depression; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive iCBT based EMI with message content, delivery frequency and timing personalised to participants' preferences.
  Interventions: Other: iCBT-based EMI
- Control group (No Intervention): Receive general mental health information through instant message.

INTERVENTIONS:
Other: iCBT-based EMI — Consists of brief iCBT for psychological support (mandatory), stroke care education (optional), and nurse-led real-time chat-based support messages, delivered according to participants' preferences.
  Arms: Intervention group

SUMMARY:
Around one third of stroke survivors develop depression at any point of time following the stroke event. Post-stroke depression (PSD) is associated with negative care outcomes including poorer function, longer hospital stays, increased outpatient and inpatient clinic use, and higher mortality rate. In Hong Kong (HK), the prevalence of PSD within the hospital setting was 36%, and up to 68% in the community setting. However, PSD is seldom addressed in either settings in HK and elsewhere. Meta-analyses reported the effectiveness of Internet-based cognitive behavioural therapy (iCBT), particularly when guided by therapists (d = 0.63). Personalised and synchronous instant message-based intervention guided by therapists is an emerging form of psychological intervention. While such intervention showed medium to large effect (Hedges' g = 0.73) on negative psychological distress episodes including depression, no study has investigated its effect on PSD. The proposed study aims to 1) investigate the effect of therapist-guided brief iCBT delivery through instant messaging applications (e.g. WhatsApp and WeChat) to provide personalised and synchronous PSD support and 2) understand the experience of and compliance with the intervention. 160 community-dwelling stroke survivors with Patient Health Questionnaire-9 (PHQ-9) scores ranging from 5 to 19 indicating mild to moderate depressive symptoms will be recruited and then individually randomised into the Intervention group (n=80) or Control group (n=80). Intervention group will receive 1) instant message-delivered brief iCBT for 3 months at participants' chosen times and frequencies, and 2) therapist-led text or voice message-based PSD support to enhance the effects of iCBT through real-time counselling and practical advice. Control group will only receive messages on general mental health information and reminders to participate in follow-up surveys. The primary outcome is PHQ-9 score at 6 months. Secondary outcomes will include anxiety (GAD-7), perceived stress (PSS-4), loneliness (ULS-8), and quality of life (EQ-5D-5L) at 6 months. The study will strictly follow the CONSORT-EHEALTH checklist. Post-trial qualitative study will be conducted to understand the participants' experience of and compliance with the intervention (n≈20) respectively. This study will provide the first and practical evidence on the effectiveness of instant message-delivered brief iCBT intervention in addressing PSD in HK and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke (ICD-10 codes: I60-I69);
* Aged ≥18;
* Able to read and communicate in Chinese (Cantonese or Putonghua);
* Able to use the text or voice messaging function on smartphone;
* MoCA 5-minute Protocol (cognitive screen) ≥14;
* Community-dwelling
* Less than 1 year after stroke event;
* PHQ-9 (depressive symptom) score ranging from 5 to 19 (note. mild: 5-9, moderate: 10-14, moderately severe: 15-19 and severe: 20-27)

Exclusion Criteria:

* Diagnosis of psychiatric disease before stroke event or currently taking psychotropic drug including antidepressants
* PHQ-9 ≥ 20 (i.e., severe depressive symptom)
* Currently participating in any type of psychological intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]) | 24-week
  A 9-item scale with score ranging from 0 to 27, higher scores indicate higher severity of depressive symptom

SECONDARY OUTCOMES:
Anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | 24-week
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptoms
Stress level (Perceived Stress Scale [PSS-4]) | 24-week
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of stress
Quality of life (EuroQol 5-dimension 5-level questionnaire [EQ-5D-5L]) | 24-week
  A 5-item scale with predicted values ranging from -.864 to 1, higher values indicate higher health-related quality of life
Loneliness level (UCLA Loneliness Scale [ULS-8]) | 24-week
  The total score (8 items) ranges from 8 to 32 points, with higher scores suggesting a higher degree of loneliness

CONTACTS AND LOCATIONS:
Locations (7):
- Hong Kong (7):
  - Hong Kong PHAB Association, Hong Kong
  - Hong Kong Stroke Association, Hong Kong
  - NT West Community Rehabilitation Day Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Hong Kong Society for Rehabilitation, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No